CLINICAL TRIAL: NCT02081690
Title: A Multi-center, Open-label, Single-arm, Phase 3b Study of Macitentan in Patients With Pulmonary Arterial Hypertension to Psychometrically Validate the French, Italian and Spanish Versions of the PAH-SYMPACT™
Brief Title: A Pulmonary Arterial Hypertension Study With Macitentan to Validate the PAH-SYMPACT™ in France, Italy and Spain
Acronym: ORCHESTRA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-055-310
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Results first posted 2018-02-05 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: PAH-SYMPACT; psychometric instrument
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Macitentan (Experimental): Macitentan tablet, dose of 10 mg, once daily
  Interventions: Drug: Macitentan

INTERVENTIONS:
Drug: Macitentan — Macitentan tablet, dose of 10 mg, once daily

SUMMARY:
Prospective, multi-center, open-label, single-arm, Phase 3b psychometric validation study.

Primary objectives: To evaluate the psychometric characteristics of reliability and construct validity of the French, Italian and Spanish versions of the PAH-SYMPACT™.

To evaluate the ability of the French, Italian and Spanish versions of the PAH SYMPACT™ to detect change.

Secondary objective: To assess the safety of macitentan in patients with pulmonary arterial hypertension (PAH).

Exploratory objective: To explore the effects of macitentan on PAH symptoms and their impact (as measured by the PAH-SYMPACT™) in patients with PAH in France, Italy and Spain.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study-mandated procedure.
2. Patients with symptomatic PAH in WHO Functional Class (FC) II or III.
3. Patients with PAH belonging to one of the following subgroups of the Dana Point Clinical Classification Group 1:

   1. Idiopathic, or,
   2. Heritable, or,
   3. Drug or toxin induced, or,
   4. Associated with one of the following:

   i. Connective tissue disease, ii. Congenital heart disease with simple systemic-to-pulmonary shunt at least 1 year after surgical repair, iii. HIV infection.
4. Documented hemodynamic diagnosis of PAH by right heart catheterization - performed at any time prior to Screening showing:

   1. Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and,
   2. Resting pulmonary vascular resitance (PVR) > 240 dyn.s.cm-5 and,
   3. Pulmonary capillary wede pressure (PCWP) or left ventricular end diastolic pressure (LVEDP) ≤ 15 mmHg.
5. 6-minute walk distance (6MWD) ≥ 150 m at Screening.
6. Able to fluently speak and read the local language.
7. Men or women aged 18-80; women of childbearing potential (as defined below) must:

   1. Have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline and agree to perform monthly serum pregnancy tests, and,
   2. Agree to use two reliable methods of contraception in parallel, from Screening Visit 1 until 1 month after study drug discontinuation (see details below).

      * A female is considered to have childbearing potential unless she meets at least one of the following criteria:

        * Previous bilateral salpingo and/or oophorectomy, or hysterectomy.
        * Premature ovarian failure confirmed by a specialist.
        * Pre-pubescence, XY genotype, Turner syndrome, uterine agenesis.
        * Postmenopausal, defined as 12 consecutive months with no menses without an alternative medical cause.
      * Of the two contraceptive methods that must be used, one must be from Group 1, and one must be from Group 2, defined as follows:

        * Group 1: Oral, implantable, transdermal or injectable hormonal contraceptives, intrauterine devices, female sterilization (tubal ligation or non surgical sterilization, e.g., permanent contraception with Essure procedure), or partner's sterilization (vasectomy). If a hormonal contraceptive is chosen from this group, it must be taken for at least 1 month prior to enrollment. Alternatively, if the Essure procedure is chosen as a contraceptive method, a hysterosalpingogram must have been performed to confirm correct location of the microinserts and tubal occlusion (as per manufacturer's recommendations).
        * Group 2: Female or male condoms, diaphragm or cervical cap, any of them in combination with a spermicide.
      * Sexual abstinence, rhythm methods, or contraception by the partner alone are not considered as acceptable methods of contraception for this study.

Exclusion Criteria:

1. Known moderate-to-severe obstructive lung disease (i.e., forced expiratory volume in one second [FEV1] < 80 % of predicted, with FEV1 / forced vital capacity [FVC] < 70%) or known significant chronic lung disease diagnosed by chest imaging (e.g., interstitial lung disease, emphysema).
2. Known moderate-to-severe restrictive lung disease (i.e., total lung capacity [TLC] < 60% of predicted value).
3. Hemoglobin < 100g/L at Screening.
4. Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 3 X upper limit of the normal range (ULN) at Screening.
5. Patients undergoing dialysis.
6. Systolic blood pressure (SBP) < 90 mmHg at Screening.
7. Body weight < 40 kg at Screening.
8. Known concomitant life-threatening diseases with a life expectancy of < 12 months.
9. Treatment with ERAs within 3 months prior to Visit 2, or scheduled to receive any of these compounds, other than macitentan, during the trial.
10. Treatment with intravenous or subcutaneous prostacyclin or prostacyclin analogs within 3 months prior to Visit 2, or scheduled to receive any of these compounds during the trial.
11. Treatment with soluble guanylate cyclase stimulator (riociguat) within 3 months prior to Visit 2, or scheduled to receive riociguat during the trial.
12. Patients who changed the dose of or discontinued phosphodiesterase type-5 inhibitor (PDE5i), inhaled prostacyclin analogues, or calcium channel blockers within 3 months prior to Visit 2.
13. Initiation of diuretics within 1 week prior to the Baseline period.
14. Patients on oral diuretics in whom the dose has not been stable for at least 1 week prior to the Baseline period.
15. Treatment with cytochrome P4500 (CYP) 3A inducers within 4 weeks prior to Visit 2.
16. Recently started (< 8 weeks prior to Visit 2) or planned cardio-pulmonary rehabilitation program based on exercise.
17. Females who are lactating or pregnant (positive Screening or Baseline pregnancy test) or plan to become pregnant during the study.
18. Known hypersensitivity to macitentan or its excipients or drugs of the same class.
19. Treatment with another investigational drug within 3 months prior to Visit 2.
20. Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as drug or alcohol dependence or psychiatric disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-10-01 (Actual); Study Completion 2015-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Loïc Perchene, Study Director — Actelion
Locations (39):
- France (13):
  - Hôpital de Haut Levêque, Bordeaux
  - Hôpital Côte de Nacre, Caen
  - Hôpital Albert Michallon, Grenoble
  - CHU de Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille - Hôpital Cardiologique, Lille
  - Hôpital Louis Pradel, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpitaux de Brabois, Nancy
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Nord, Saint-Etienne
  - Hôpital Civil, Strasbourg
  - Hôpital Larrey, Toulouse
- Italy (12):
  - Universita degli Studi di Bari, Bari
  - Ospedale di Venere, Bari
  - Ospedale Sant'Orsola, Bologna
  - A.O.U.C. Careggi, Florence
  - Milan Sacco Hospital, Milan
  - AORN Azienda Ospedaliera dei Colli, Naples
  - Ambulatorio Scompenso Cardiaco e Trapiant, Pavia
  - Istituto di Fisiologia clinica - CNR, Pisa
  - Centro Per La Diagnosi E La Cura Dell'Ipertensione Polmonare, Roma
  - UOC Immunologia Clinica B-PGRM Centro di Riferimento per la Sclerosi Sistemica, Rome
  - Ospedale "S. Maria di Cà Foncello", Treviso
  - Policlinico G.B. Rossi, Verona
- Spain (14):
  - Hospital Universitario Insular Gran Canarias, Las Palmas de Gran Canaria, Canary Islands
  - Hospital General de Alicante, Alicante
  - Hospital Val Hebron, Barcelona
  - Hospital Clinic, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Reina Sofia, Córdoba
  - Hospital Dr Negrin, Las Palmas de Gran Canaria
  - Hospital 12 Octubre, Madrid
  - Hospital La Paz, Madrid
  - Hospital Carlos Haya, Málaga
  - Hospital Son Espases, Palma de Mallorca
  - Hospital de Valdecilla, Santander
  - Hospital Virgen del Rocio, Seville
  - Hospita General U. Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was designed to recruit 160 male and female patients aged 18 to 80 years (inclusive) with PAH. A total of 93 patients were screened and 88 patients were enrolled at 37 recruitment sites. Due to slow recruitment, the sponsor decided to prematurely stop the study.
Groups:
- Macitentan: Subjects received Macitentan at a 10 mg oral dose, once daily during 16 weeks
Period: Overall Study
Arm/Group | Macitentan
Started | 88
Completed | 81
Not Completed | 7
Not completed — Death | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Macitentan
Number analyzed (Participants) | 88
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 57.5 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Reliability and the Construct Validity of the Cardiopulmonary Symptoms Domain of the PAH-SYMPACT
Description: The Cardiopulmonary Symptoms domain consists of 6 items reported on a 5-point Likert scale (from 0 to 4). The value 0 means "no symptom" and value 4 corresponds to "very severe symptoms".The symptoms part of the PAH-SYMPACT was administered daily over a 7 day period. The recall period of symptom items is the last 24 hours. An average Cardiopulmonary Symptoms domain score is determined based on the daily scores of the 6 items. It was administered two times (daily during 7 days each time) prior to administration of Macitentan (Visit 2, Baseline) and daily during the 7-day period in the treatment period prior to Visit 3 (Week 8) and Visit 4 (Week 16).
Time Frame: From Screening Visit (Visit 1) to End of Treatment (EOT) Visit (Visit 4, Week 16)
Population: Validation set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 87
Score on a scale
  Cardiopulmonary Symptoms domain score at baseline | 0.90 (0.58)
  Cardiopulmonary Symptoms domain score at week 8 | 0.89 (0.63)
  Cardiopulmonary Symptoms domain score at week 16 | 0.89 (0.68)

2. Primary Outcome: Evaluation of the Reliability and the Construct Validity of the Cardiovascular Symptoms Domain of the PAH-SYMPACT
Description: The Cardiovascular Symptoms domain consists of 5 items reported on a 5-point Likert scale (from 0 to 4). The value 0 corresponds to "no symptoms" and value 4 corresponds to "very severe symptoms". The symptoms part of the PAH-SYMPACT was administered daily over a 7 day period. The recall period of symptom items is the last 24 hours. An average Cardiovascular Symptoms domain score is determined based on the daily scores of the 5 items. It was administered two times (daily during 7 days each time) prior to administration of Macitentan (Visit 2, Baseline) and daily during the 7-day period in the treatment period prior to Visit 3 (Week 8) and Visit 4 (Week 16).
Time Frame: From Screening Visit (Visit 1) to End of Treatment (EOT) Visit (Visit 4, Week 16)
Population: Validation set
Measure: Median (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 87
Score on a scale
  Cardiovascular Symptoms domain score at baseline | 0.58 (0.62)
  Cardiovascular Symptoms domain score at week 8 | 0.54 (0.62)
  Cardiovascular Symptoms domain score at week 16 | 0.54 (0.65)

3. Primary Outcome: Evaluation of the Reliability and the Construct Validity of the Physical Impacts Domain of the PAH-SYMPACT
Description: The Physical Impacts domain consists of 7 items reported on a 5-point Likert scale (from 0 to 4). The value 0 corresponds to "not at all"/"with no difficulty at all" and value 4 corresponds to "very much"/"extremely"/ "not able at all". The impacts part of the PAH-SYMACT was administered on Day 7 of the symptoms part administration. Items in the impact part have a 7 day recall period. An average Physical Impacts domain score is determined based on the 7 items in the domain. It was administered two times prior to administration of Macitentan (Visit 2, Baseline) and during the 7-day period in the treatment period prior to Visit 3 (Week 8) and Visit 4 (Week 16).
Time Frame: From Screening Visit (Visit 1) to End of Treatment (EOT) Visit (Visit 4, Week 16)
Population: Validation set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 87
Score on a scale
  Physical Impacts domain score at baseline | 1.13 (0.88)
  Physical Impacts domain score at week 8 | 1.15 (0.97)
  Physical Impacts domain score at week 16 | 1.25 (1.00)

4. Primary Outcome: Evaluation of the Reliability and the Construct Validity of the Cognitive/Emotional Impacts Domain of the PAH-SYMPACT
Description: The Cognitive/Emotional Impacts domain consists of 4 items reported on a 5-point Likert scale (from 0 to 4). The value 0 corresponds to "not at all"/"with no difficulty at all" and value 4 corresponds to "very much"/"extremely"/ "not able at all". The impacts part of the PAH-SYMACT was administered on Day 7 of the symptoms part administration. Items in the impact part have a 7 day recall period. An average Cognitive/Emotional Impacts domain score is determined based on the 4 items in the domain. It was administered two times prior to administration of Macitentan (Visit 2, Baseline) and during the 7-day period in the treatment period prior to Visit 3 (Week 8) and Visit 4 (Week 16)."
Time Frame: From Screening Visit (Visit 1) to End of Treatment (EOT) Visit (Visit 4, Week 16)
Population: Validation set
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Macitentan
Number analyzed (Participants) | 83
Score on a scale
  Cogn/Emotional Impacts domain score at baseline | 0.87 (0.77)
  Cogn/Emotional Impacts domain score at week 8 | 0.88 (0.91)
  Cogn/Emotional Impacts domain score at week 16 | 0.91 (0.96)

ADVERSE EVENTS:
Time Frame: From study treatment initiation up to 30 days after study treatment discontinuation
Arm/Group | Macitentan
All-Cause Mortality (participants affected / at risk) | 3/88
Serious Adverse Events (participants affected / at risk) | 13/88
Other Adverse Events (participants affected / at risk) | 21/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=88)
Arteriovenous fistula (Vascular disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Investigation (Investigations) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Right ventricular failure (Cardiac disorders) | 4 (5)
Sympathectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Macitentan (N=88)
Headache (Nervous system disorders) | 11 (12)
Hypotension (Vascular disorders) | 5 (6)
Oedema peripheral (General disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study-related publication written independently by investigators must be submitted to Actelion for review at least 30 days prior to submission for publication or presentation. Upon review, Actelion may provide comments, and may also request alterations and/or deletions for the sole purpose of protecting its confidential information and/or patent rights.